CLINICAL TRIAL: NCT02876978
Title: Preliminary Clinical Study of Autologous T Cells Modified Chimeric Antigen Receptor (CAR) Targeting GPC3 for the Treatment of Recurrent or Refractory Lung Squamous Cell Carcinoma
Brief Title: Anti-GPC3 CAR T for Recurrent or Refractory Lung Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG1003
Record Dates: First submitted 2016-08-09; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Lung Squamous Cell Carcinoma
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAR-GPC3 T cells (Experimental): Intravenous infusion with escalating dose is adopted in this study.
  Total dosage: 1 x 10^5 - 2 x 10^9 CAR-GPC3 T cells/kg
  The next dose and interval depends on the response of the subject to previous dose.
  Lymphodepletion:
  Fludarabine: 30 mg/m^2/day x 4 days; Cyclophosphamide: 500 mg/m^2/day x 2 days. Adjustment is in discretion of the investigator based on individual response.
  Interventions: Genetic: CAR-GPC3 T Cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: CAR-GPC3 T Cells — Intravenous infusion of CAR-GPC3 T cells is conducted 1 - 2 days following lymphodepletion.
  Other Names: Anti-GPC3 CAR T; CAR T cells redirected to Glypican-3
Drug: Fludarabine — 30 mg/m^2/day x 4 days
Drug: Cyclophosphamide — 500 mg/m^2/day x 2 days

SUMMARY:
The purpose of this study is to observe and confirm the safety, tolerance and cell pharmacokinetics of lentivirus-transduced CAR-GPC3 T cells (CAR-GPC3 T cells targeting GPC3)

DETAILED DESCRIPTION:
A single-center, open-label pilot study to determine the safety, tolerance and engraftment potential of CAR-GPC3 T cells in subjects with GPC3+ positive lung squamous cell carcinoma.

Primary objectives:

Observe and determine the safety and tolerance in escalating dose infusion of CAR-GPC3 T cells (CAR T cells targeting GPC3) transduced with the lentiviral vector, and the survival of the CAT-GPC3 T cells in vivo, referred to as engraftment potential.

Secondary objectives:

The following indexes are monitored for curative effect of CAR-GPC3 T cells on lung squamous cell carcinoma:

1. Objective response rate (ORR), is defined as the ratio of patients diagnosed as partial remission (PR) to complete remission (CR) according to RECIST 1.1 criteria.
2. Progression free survival (PFS), is defined as the duration from baseline to PD (audited and confirmed by independent imaging), or to the day of any death event. The earlier one shall prevail.
3. Time to tumor progression (TTP), is defined as the duration from baseline to disease starts to get worse or spreads to other parts of the body.
4. Overall survival (OS), is defined as the time period from the 1st day of treatment to the day of death for any reason. For patients who are still alive at the data analysis day, OS data is subject to the last confirmed time of survival patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18~70 years old
2. Subjects are diagnosed as refractory, recurrent ,metastatic, advanced lung squamous cell carcinoma by histological and cytological methods including specific lesion-targeted brush biopsy, lavage and fine needle aspiration;
3. Have at least one new measurable tumor lesion compared with previous irradiated region
4. Tumor tissues samples confirmed as GPC3-positive
5. Expected survival≥12 weeks
6. ECOG scored as 0-1 or KPS grading > 80
7. ANC≥1500/nm3
8. PLT≥100000/mm3
9. Hb≥9.0g/dL
10. Serum creatinine≤2.5mg/dL，CCR≥50ml/min (renal malfunction defined as CCR<50ml/min according to Cockroft-Gault formula)
11. ALT and AST≤2.5ULN; for liver metastasis，ALT and AST ≤5ULN
12. Serum TBiL≤3.0mg/dL, TBiL≤2.5ULN
13. PT: INR < 1.7 or extended PT to normal value < 4s
14. Adequate venous access for apheresis or venous blood collection, and no other contraindication of blood cell separation
15. Patients with willingness to be in this study and able to provide informed consent
16. Capable of receiving treatment and follow up, included subjects are required to receive treatment in the enrolled centre
17. Women of childbearing age are required to take acceptable measures to minimize the possibility of pregnancy during whole session. Women of childbearing age must have negative results of serum or urine tests within 24 hours prior to infusion. Women subjects must not be in lactation;

Exclusion Criteria:

1. CAR-T positive rate < 10%
2. pregnant women or women in lactation
3. active HBV or HCV infection
4. HIV/AIDS infection
5. active infection
6. previously suffered from diseases or concurrent diseases as followed：

   * patients confirmed as severe autoimmune diseases in long-term (over 2 months) need of systemic immune inhibitors (steroid) or as immune-mediated symptomatic diseases including ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE), autoimmune vasculitis (for example, Wegener's granulomatosis)
   * subjects with previous diagnosis as motor neurone disease caused by autoimmunity
   * subjects previously suffered from toxic epidermal necrolysis (TEN)
   * subjects with any mental diseases including dementia, mental status change that may impinge the understanding and performance of informed consent and related questionnaire
   * subjects with severe, uncontrollable diseases judged by investigators that may hinder them receiving this treatment
   * subjects with previously active malignant tumors including basal or squamous skin cancer, superficial bladder cancer, and in situ breast carcinoma within 5 years who had been completely cured without the need of follow-up treatment are not excluded.
7. during ongoing treatment using systemic steroid or steroid inhalants
8. previous treatment used gene therapy products
9. previous experience of immunotherapies including CIK, DC, DC-CIK, LAK for the treatment of cancer
10. allergic to immunotherapies or related drugs
11. patients in need of treatment for heart disease with ≥2 NYHA or for poor controlled hypertension
12. subjects with unstable or active peptic ulcer or alimentary tract hemorrhage
13. subjects with previous organ transplantation or ready for organ transplantation
14. subjects in need of anticoagulant therapy treatment (warfarin or heparin)
15. subjects judged by investigators as not appropriate for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance: Occurrence of study related adverse events | 24 weeks
  Occurrence of study related adverse events, defined as laboratory toxicities and clinical events that are possibly, likely or definitely related to study treatment at any time from the infusion until week 24. This will include infusive toxicity, and any toxicity possibly related to the CAR-GPC3 T cells.

SECONDARY OUTCOMES:
Engraftment: the DNA vector copies per mL blood of CAR-GPC3 T cells | 2 years
  The DNA vector copies per mL blood of CAR-GPC3 T cells on week 4 after the first infusion by Q-PCR. Q-PCR for CAR-GPC3 vector sequences will also be performed after infusion thereafter until any 2 sequential tests are negative documenting loss of CAR-GPC3 T cells within 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Liyan, MD, Principal Investigator — Shanghai Chest Hospital,Shanghai Jiaotong University
Locations (1):
- Shanghai Chest Hospital,Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No